CLINICAL TRIAL: NCT06546020
Title: PARTNERSHIP: Elucidating Gut Microbiota-dependent Health Impacts of Haskap Berries to Inform Agricultural Production Practices That Will Maximize Bioactive Potential
Brief Title: Gut Microbiota-dependent Health Impacts of Haskap Berries
Acronym: HIH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montana State University (Other)
Collaborators: Montana State Agricultural Experiment Station (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2024-1417-FCR
Record Dates: First submitted 2024-08-01; First posted 2024-08-09 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Metabolic Disease; Inflammation; Microbial Colonization
Keywords: Microbial metabolism; Gut microbial composition; Serum metabolome; Polyphenols
MeSH Terms: conditions — Metabolic Diseases; Inflammation; Communicable Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Placebo and haskap interventions were designed to be comparable in taste and appearance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo, Metabolically Healthy (Placebo Comparator): The placebo supplement will have no polyphenol content and will be carbohydrate-matched to the experimental group. A twice daily dose (10-12 hours apart) will be consumed for 8 weeks.
  Interventions: Dietary Supplement: Placebo comparator
- Haskap, Metabolically Healthy (Experimental): The haskap supplement will consist of a haskap berry smoothie. A twice daily dose (10-12) hours apart will be consumed for 8 weeks.
  Interventions: Dietary Supplement: Haskap berry smoothie
- Placebo, Metabolically Unhealthy (Placebo Comparator): The placebo supplement will have no polyphenol content and will be carbohydrate-matched to the experimental group. A twice daily dose (10-12 hours apart) will be consumed for 8 weeks.
  Interventions: Dietary Supplement: Placebo comparator
- Haskap, Metabolically Unhealthy (Experimental): The haskap supplement will consist of a haskap berry smoothie. A twice daily dose (10-12) hours apart will be consumed for 8 weeks.
  Interventions: Dietary Supplement: Haskap berry smoothie

INTERVENTIONS:
Dietary Supplement: Haskap berry smoothie — A smoothie blend of berries and water
  Arms: Haskap, Metabolically Healthy; Haskap, Metabolically Unhealthy
Dietary Supplement: Placebo comparator — A smoothie with no polyphenolic content and matched in carbohydrate composition to the experimental haskap smoothie
  Arms: Placebo, Metabolically Healthy; Placebo, Metabolically Unhealthy

SUMMARY:
Polyphenol-rich Haskap berries (Haskap) have untapped therapeutic potential to improve human health, and agricultural producers in northern U.S. states are poised to increase production if consumer demand increases. A critical knowledge gap is that little is known about the interactions between gut microbes and Haskap polyphenols to produce bioactive metabolites linked to downstream health impacts. Additionally, little is known about which Haskap varieties and harvest timing yield the greatest bioactive potential. This study aims to address these gaps by investigating the interaction of bioactive components in Haskap with gut microbiota and the resultant gut and serum metabolites, inflammation, and metabolic health, and then couple this with analysis of berries from different Haskap varieties and harvest times.

DETAILED DESCRIPTION:
The long-term goal of this project is to form a partnership linking the health impacts of Haskap varieties and management practices that maximize health-promoting compounds to benefit both consumers and producers. Specific objectives of this study are to determine 1) the impact of Haskap on the gut microbiome and metabolome, 2) how gut microbiome composition and production of bioactive metabolites from Haskap impacts health and inflammation biomarkers, and 3) which Haskap varieties and growing practices increase production of health-promoting compounds.

To accomplish this, a four-armed, randomized, triple-blind, placebo controlled clinical trial of Haskap versus placebo for two separate groups with distinctly low and high metabolic syndrome status will be completed. Participants will be assessed for health biometrics, fat oxidation, gut microbiome composition, inflammation, and both the gut and serum metabolome before and after 8 weeks of intervention. Haskap fruit from twenty varieties will primarily come from the randomized block design field trial and fruit will be harvested at four stages of fruit maturity, then analyzed for polyphenol content. This part of the study will be replicated over three growing seasons.

ELIGIBILITY:
Inclusion Criteria for Metabolically Healthy Group:

All of the following:

* Waist circumference: men ≤ 40, women ≤ 35 inches
* Systolic blood pressure: ≤ 130 mmHg
* Diastolic blood pressure: ≤ 85 mmHg
* Fasting glucose: ≤ 100 mg·dl-1
* Fasting triglycerides: ≤ 150 mg·dl-1
* HDL: men > 40, women > 50 mg·dl-1

Inclusion Criteria for Metabolically Unhealthy Group:

Required:

- Waist circumference: men ≥ 40, women ≥ 35 inches

AND ≥ 1 of the following:

* Systolic blood pressure: > 130 mmHg
* Diastolic blood pressure: > 85 mmHg
* Fasting glucose: > 100 mg·dl-1
* Fasting triglycerides: > 150 mg·dl-1
* HDL: men ≤ 40, women ≤ 50 mg·dl-1

Exclusion Criteria:

* BMI <18 or > 40 kg/m^2
* potential allergy to Haskap or placebo ingredients
* use of anti-inflammatory, lipid lowering, glucose lowering, blood pressure, or any other medications that may interfere with study measures
* pregnant or lactating woman
* diagnosis with type 1 or type 2 diabetes or any other condition that may interfere with study measures
* smoke cigarettes
* have taken antibiotics in the past 90 days
* take supplements including pre/probiotics or "superfoods" within 30 days of starting the study
* are planning on starting a weight loss or exercise regiment change
* follow a specific diet such as low carbohydrate, vegan, and vegetarian
* consume over 5 servings of fruit/vegetables per day
* are unwilling to reduce caffeine intake to one 8 oz serving per day for the durations of the study

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
16 subunit ribosomal ribonucleic acid (16S rRNA) gut microbial composition | 8 weeks
  fecal microbial composition
Inflammation (pg/mL) | 8 weeks
  Serum interleukin (IL) IL-1B, IL-6, IL-10, IL-17, IL-23, tumor necrosis factor alpha (TNF-alpha), granulocyte-macrophage colony-stimulating factor (GM-CSF), interferon gamma (IFN-gamma)
Lipid Panel (mg/dL) | 8 weeks
  Serum triglycerides (TG), low-density lipoprotein (LDL) cholesterol, high-density lipoprotein (HDL) cholesterol, total cholesterol (CHOL), glucose (GLU)
F2 isoprostanes | 8 weeks
  urine
Untargeted metabolomic analysis | 8 weeks
  Serum metabolome
Untargeted metabolomic analysis | 8 weeks
  Fecal metabolome
Exercise Induced Fat Oxidation | 8 weeks
  Measurement in g/min of fat being utilized during exercise at 40-60% of the participants estimated VO2max

SECONDARY OUTCOMES:
Acute Diet | 8 weeks
  24-hour dietary recall using the Automated Self-Administered 24-hour Dietary. Assessment Tool (ASA24). Outcome is macronutrient and micronutrient composition of food entry.
Habitual Diet | Baseline
  Habitual diet recall using Dietary History Questionnaire (DHQ) III (1 year recall). Outcome measures are healthy eating index (HEI) scores which include nine components based on adequacy (total fruit, whole fruit, total vegetables, greens and beans, whole grains, dairy, total protein foods, seafood and plant proteins, fatty acids) and four components based on moderation (refined grains, so-dium, added sugars, saturated fats). Each component is ranked 1-10 in order of increasing health. Total HEI score is reported as the sum of all components (100 possible points) with more points indicating increased health of diet.
Anthropometric Assessments | 8 weeks
  waist circumference (cm)
Anthropometric Assessments | 8 weeks
  visceral adipose (L)
Anthropometric Assessments | 8 weeks
  BMI (kg/m2)
Anthropometric Assessments | 8 weeks
  fat free mass (%)
Blood pressure | 8 weeks
  SBP/DBP (mmHG)
Estimated VO2 max | 0 weeks
  Estimation of participants VO2 max (ml/k/min) from a Fatmax test

CONTACTS AND LOCATIONS:
Overall Officials: Mary P Miles, PhD, Principal Investigator — Montana State University
Locations (1):
- Montana State University, Bozeman, Montana, United States

DOCUMENTS (3):
  • Study Protocol (2024-11-05): https://cdn.clinicaltrials.gov/large-docs/20/NCT06546020/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-05): https://cdn.clinicaltrials.gov/large-docs/20/NCT06546020/SAP_001.pdf
  • Informed Consent Form (2024-11-05): https://cdn.clinicaltrials.gov/large-docs/20/NCT06546020/ICF_002.pdf